CLINICAL TRIAL: NCT06494371
Title: An Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of CD30-Targeted LCAR-HL30 Cells in Patients With Relapsed/Refractory Hodgkin's Lymphoma and Anaplastic Large Cell Lymphoma
Brief Title: A Study of LCAR-HL30 in Subjects With Relapsed/Refractory Hodgkin's Lymphoma and Anaplastic Large Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2203-0001
Record Dates: First submitted 2024-06-18; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Hodgkin's Lymphoma; Anaplastic Large Cell Lymphoma
Keywords: Hodgkin's Lymphoma; Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor T cells LCAR-HL30 cells (Experimental): Each subject will receive LCAR-HL30 cells.
  Interventions: Biological: LCAR-HL30 cells

INTERVENTIONS:
Biological: LCAR-HL30 cells — Prior to infusion of the LCAR-HL30, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine

SUMMARY:
This is a prospective, single-arm, open-label, exploratory clinical study of LCAR-HL30 in adult subjects with relapsed/refractory Hodgkin's Lymphoma and Anaplastic Large Cell Lymphoma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label exploratory clinical study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor efficacy profiles of LCAR-HL30, a chimeric antigen receptor(CAR)-T cell therapy in subjects with relapsed/refractory Hodgkin's Lymphoma and Anaplastic Large Cell Lymphoma. Patients who meet the eligibility criteria will receive LCAR-HL30 infusion. The study will include the following sequential stages: screening, pre-treatment (cell product preparation: lymphodepleting chemotherapy), treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical research.
2. Aged 18 to 75 years, either sex.
3. Eastern Cooperative Oncology Group (ECOG) score 0-1 (Dose escalation phase). ECOG score 0-2 (Dose expansion period).
4. Histologically confirmed Hodgkin's lymphoma or Anaplastic large cell lymphoma with positive CD30 expression.
5. At least one evaluable tumor lesion according to Lugano 2014 criteria.
6. Expected survival ≥3 months.
7. Clinical laboratory values in the screening period meet criteria.
8. Effective contraception.

Exclusion Criteria:

1. Prior antitumor therapy with insufficient washout period.
2. Previous treatment with CAR-T therapy, allogeneic hematopoietic stem cell transplantation.
3. Severe underlying diseases;
4. Hepatitis B virus surface antigen (HbsAg), Hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C virus ribonucleic acid (HCV RNA) or human immunodeficiency virus antibody (HIV-Ab) positive.
5. Presence of other serious pre-existing medical conditions that may limit patient participation in the study. Any condition that, in the investigator's judgment, will make the subject unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  An adverse event refers to any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product (investigational or non-investigational), which does not necessarily have a causal relationship with the treatment.
Pharmacokinetics in peripheral blood | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  CAR positive T cells levels in peripheral blood after LCAR-HL30 infusion.
Pharmacokinetics in peripheral blood | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  CAR transgene levels in peripheral blood after LCAR-HL30 infusion.
Pharmacokinetics in bone marrow | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  CAR positive T cells levels in bone marrow after LCAR-HL30 infusion.
Pharmacokinetics in bone marrow | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  CAR transgene levels in bone marrow after LCAR-HL30 infusion.
Recommended Phase 2 Dose (RP2D) regimen finding | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  RP2D established through accelerated titration design (ATD) and Bayesian Optimal Interval (BOIN) design.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) after administration | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  ORR is defined as the proportion of subjects who achieve complete response (CR) or partial response (PR) after treatment via LCAR-HL30 cell infusion, and the objective tumor response rate will be calculated for patients with measurable disease per the Lugano Classification for Initial Evaluation, Staging, and Response Assessment of Hodgkin and Non-Hodgkin Lymphoma (Lugano 2014).
Time to Response (TTR) after administration | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  TTR is defined as the time from the date of first infusion of LCAR-HL30 to the date of the first response evaluation of the subject who has met all criteria for PR or better.
Duration of Remission (DoR) after administration | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  DoR is defined as the time from the first documentation of remission (PR or better) to the first documented disease progression evidence (according to Lugano 2014) of the responders (who achieve PR or better response).
Progression-free Survival (PFS) after administration | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  PFS is defined as the time from the date of first infusion of the LCAR-HL30 to the first documented disease progression (according to Lugano 2014) or death (due to any cause), whichever occurs first.
Overall Survival (OS) after administration | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  OS is defined as the time from the date of first infusion of LCAR-HL30 to death of the subject.
Incidence of anti-LCAR-HL30 antibody | Minimum 2 years after LCAR-HL30 infusion (Day 1), maximum 4 years after LCAR-HL30 infusion (Day 1)
  The incidence of anti-LCAR-HL30 antibody in patients who received LCAR-HL30 infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No